CLINICAL TRIAL: NCT03868865
Title: Effects of an Integrative Day-care Clinic Program for Breast Cancer Patients During Chemotherapy: an Observational Study
Brief Title: Effects of an Integrative Day-care Clinic Program for Breast Cancer Patients During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Dr. med. Petra Voiss, Study physician, Universität Duisburg-Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-7909-BO
Record Dates: First submitted 2019-02-27; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer; Chemotherapy; Mind-Body-Medicine; Acupuncture; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative mind-body-medicine group program (Experimental): The 66 hour program encompasses mindfulness training, yoga, moderate exercise, nutrition, naturopathic self-help strategies, cognitive restructuring and acupuncture for the management of side effects caused by chemotherapy.
  Interventions: Behavioral: Integrative mind-body-medicine group program

INTERVENTIONS:
Behavioral: Integrative mind-body-medicine group program — The mind-body-medicine group program focuses on support in coping with the disease, in lifestyle modification and in reduction of chemotherapy induced side effects. The self-contained modules of the mind-body-medicine group program can be followed in an individual order, to allow adoption to different chemotherapy concepts and continued access is possible. Patients can join in the group program eleven times for six hours each visit. They participate in every one of the eleven modules once.

SUMMARY:
The aim of the study was to evaluate a new integrative day-care clinic concept for breast cancer patients receiving chemotherapy. This is an explorative pilot study. Therefore, all outcomes are analyzed exploratively.

ELIGIBILITY:
Inclusion Criteria:

* curative malignancy (breast cancer of TNM (T: primary tumor, N: regional nodes, M: metastasis) staging I-III)
* receiving chemotherapy
* at least 18 years old
* written informed consent
* willing and physically/mentally able to participate in a six hours day care clinic program eleven times during chemotherapy.

Exclusion Criteria:

* insufficient knowledge of the German language
* physical or mental disabilities resulting in ineligibility for participation in the program or filling out the questionnaires.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2015-04-07 (Actual)

PRIMARY OUTCOMES:
European Organization for Research and Treatment of Cancer (EORTC) QoL questionnaire (QLQ-C30) | up to 26 weeks (depending on chemotherapy regime)
  Besides the global quality of life subscale, this instrument assesses five functional domains of quality of life: physical, role, emotional, cognitive, and social function. Symptom scales further assess fatigue, pain, nausea and vomiting, dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial difficulties. Scores of all subscales range from 0 to 100, while a higher score represents a better level of functioning or a worse amount of symptoms.
Hospital Anxiety and Depression Scale (HADS) | up to 26 weeks (depending on chemotherapy regime)
  It measures the 2 dimensions anxiety and depression. Scores range from 0 to 21 with higher values indicate higher distress. Values of >8 indicate potential subclinical anxiety or depressive disorders
Brief Fatigue Inventory (BFI) | up to 26 weeks (depending on chemotherapy regime)
  BFI has been validated as a short and comprehensive instrument to assess severity of fatigue (three questions) and fatigue-related impairment (six questions) in cancer patients with a 9-item, 11-point rating scale. Higher scores on the BFI correspond to greater severity of fatigue / impairment through fatigue over the past 24 hours.
Perceived Stress Scale (PSS) | up to 26 weeks (depending on chemotherapy regime)
  Perceived stress was assessed by the 10-item version of the PSS, rated for the past month on a 5-point rating scale. For the summed items (range from 0 to 40) a higher total score indicates greater stress.
Satisfaction with the program | up to 26 weeks (depending on chemotherapy regime)
  Satisfaction was assessed at T1 by 5 questions regarding fulfilled expectations about the program contents, relevance for coping with cancer, social support of the group setting, transferring into everyday life, and recommendation of the program. Each question could be scored from 1=totally agree to 6=totally disagree.
Patients and numbers of adverse events | up to 26 weeks (depending on chemotherapy regime)
  All adverse events that occurred during the study period were recorded by the study physician during each day care clinic visit, regardless of their potential relation to the study intervention. After the intervention, patients were also asked to report adverse events not previously mentioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided